CLINICAL TRIAL: NCT07156318
Title: Effects of Drumming Lessons on Brain and Behavior in Children With Down Syndrome
Brief Title: Drumming Lessons' Influence on Children With Down Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Amy Needham, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 230465
Record Dates: First submitted 2025-08-15; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Down Syndrome
Keywords: Children with Down syndrome;; Effects of drumming lessons; Effects on brain and behavior; Inhibitory control; Beat perception; Intervention study
MeSH Terms: conditions — Down Syndrome; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group will receive the drumming lesson intervention between baseline and testing approximately 2 to 3 months later, so the effects of the intervention can be assessed in the lab measures.
  Interventions: Behavioral: 2 months of drumming lessons given by a professional drummer with extensive experience working with children with Down syndrome
- Control group (Other): Children in the Control condition will receive drumming lessons only after they have completed lab baseline and testing measures, about 2 to 3 months later.
  Interventions: Behavioral: Lessons after measurement

INTERVENTIONS:
Behavioral: 2 months of drumming lessons given by a professional drummer with extensive experience working with children with Down syndrome — Drumming lessons consisting of how to use hands to drum on djembe drum, using alternating hands to drum, drumming to a metronome and to music.
  Arms: Experimental group
Behavioral: Lessons after measurement — Receiving lessons after the two lab visits should still offer any possible positive effects to participants while still allowing us to compare the Control group children's behaviors to those of the Experimental group.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if drumming lessons can increase self-control in children with Down syndrome. The main question it aims to answer is whether 2 months of drumming lessons can improve the behavioral control and timing skills in children with Down syndrome. Participants are between 7 and 15 years of age and receive two months of drumming lessons given by a professional drummer with extensive experience working with children with Down syndrome. Children in the experimental group visit our lab once before lessons start and once after lessons are completed. Children in the control group visit our lab twice before they start their lessons. Lab visits include brain recordings taken using a net-style cap, computer tasks, and drumming to music.

DETAILED DESCRIPTION:
Down syndrome (DS) is the most common chromosomal cause of cognitive disability, and it affects approximately 1 in 700 live births. Although the genetic etiology of DS (a complete or partial third 21st chromosome) has been known for over 50 years, many fundamental questions about how to support high quality of life for individuals with DS remain unanswered. One area of relative weakness in DS is Inhibitory Control (IC). This skill is important for daily tasks such as following directions, making decisions, and managing money among other tasks. Existing research demonstrates a clear link between playing the drums and IC. In the proposed research, we will conduct an experiment in which 7- to 12-year-old children are randomly assigned to the Experimental (EXP) and Wait List Control (WLC) conditions. In the EXP condition, children will receive drumming lessons between Visit 1 and Visit 2, and in the Wait List Control group, children will receive drumming lessons after Visit 2. In this way, all children will receive drumming lessons, but only the EXP group will show effects of the drumming lessons in Visit 2. Testing conducted during Visits 1 and 2 will include behavioral and neural measures of inhibitory control and drumming, neural measures of beat perception, and parent report of social behavior (via Standardized questionnaire). Our predictions are that children in the EXP condition will show improvements in both measures of IC and increases in precision in the beat perception and drumming tasks. We also expect that parent report of children's behavior on the social skills questionnaire will show improvement. Across the EXP and WLC conditions, we expect no differences at Visit 1 but significant differences between conditions at Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome

Exclusion Criteria:

* Already taken drumming lessons
* Uncorrected hearing loss
* Uncorrected vision loss

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Zoo task | Baseline to two months
  Behavioral "Go/No go" task done on a computer designed to assess children's inhibitory control
Statue task | Baseline to two months
  Child is encouraged to 'become a statue' by holding their body in a position and not moving
Beat Perception | Baseline to two months
  EEG measure of brain activity during passive listening to music
Beat production | Baseline to two months
  EEG and behavioral measures of when child thinks beat is happening during music or metronome

CONTACTS AND LOCATIONS:
Overall Officials: Amy Needham, PhD, Principal Investigator — Vanderbilt University; Miriam Lense, PhD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
In this initial investigation, it seems unlikely that data at the participant level would be informative to other researchers. If it becomes clear during the study that sharing of IPD actually would be beneficial, we will recontact participants for their consent to share this information and share those datasets for which we obtain consent.

REFERENCES:
- [Background] Cahart MS, Amad A, Draper SB, Lowry RG, Marino L, Carey C, Ginestet CE, Smith MS, Williams SCR. The effect of learning to drum on behavior and brain function in autistic adolescents. Proc Natl Acad Sci U S A. 2022 Jun 7;119(23):e2106244119. doi: 10.1073/pnas.2106244119. Epub 2022 May 31. PMID 35639696